CLINICAL TRIAL: NCT05287685
Title: Adapting a Parenting Intervention to Promote Healthy Screen Time Habits in Young Children With Externalizing Behavior Problems
Brief Title: Adapting a Parenting Intervention to Promote Healthy Screen Time Habits in Young Children With Behavior Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21HD104367-01A1 (NIH); 1R21HD104367-01A1 (NIH)
Record Dates: First submitted 2022-02-22; First posted 2022-03-18 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Behavior Problem; Parenting
Keywords: child screen media use; behavior; parenting
MeSH Terms: conditions — Mental Disorders; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Teachers rating behavior and independent coders assessing parent-child interactions will be masked to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screen media adapted School Readiness Parenting Program (Experimental): Screen media adapted School Readiness Parenting Program (Once weekly session of 1.5 hours for 8 weeks)
  Interventions: Behavioral: Screen media adapted School Readiness Parenting Program
- Original School Readiness Parenting Program (Active Comparator): Original School Readiness Parenting Program (Once weekly session of 1.5 hours for 8 weeks)
  Interventions: Behavioral: School Readiness Parenting Program

INTERVENTIONS:
Behavioral: Screen media adapted School Readiness Parenting Program — For the screen time adapted parenting intervention, screen time intervention components will be infused into the SRPP (described below) to address three primary areas shown in research to play an important role in healthy screen media use: (1) reducing and managing screen time use; (2) maximizing benefits of screen time content; and (3) promoting positive parent-child interactions during co-use of screen media. Psychoeducation and practice of these strategies will be incorporated into sessions of the SRPP in which relevant behavioral concepts are addressed.The screen time adapted parenting intervention will utilize the same format (large group, 8 weekly 1.5 hour sessions) as the SRPP.
  Arms: Screen media adapted School Readiness Parenting Program
Behavioral: School Readiness Parenting Program — The SRPP is an 8-week parenting program for parents of preschool aged children with externalizing behavior problems. The SRPP targets child externalizing behavior problems specifically, as well as to help parents promote children's school readiness skills. The SRPP follows a group Parent-Child Interaction Therapy (PCIT) model and also uses motivational interviewing and modelling problem solving approaches. The SRPP utilizes a large group format (10-15 parents) with weekly sessions lasting 1.5 hours. The SRPP curriculum contains traditional aspects of behavioral management strategies (e.g., improving parenting skills and the parent-child relationship; discipline strategies such as time out). Specific sessions of the SRPP also directly target parental interactions during children's learning activities and setting up homework and household structure and routines. In its original form, SRPP does not address children's screen time.
  Arms: Original School Readiness Parenting Program

SUMMARY:
This project is a study funded by the National Institute of Child Health and Human Development to develop and pilot test an adapted parenting intervention to decrease excessive/inappropriate screen media use in young children with externalizing behavior problems.

DETAILED DESCRIPTION:
The goal of this study is to develop and pilot test an adapted screen time intervention for parents of young children with externalizing behavior problems. As young children's access and exposure to different types of screen media devices has increased, so has public health concern around the links between unhealthy early screen media use (including excessive use and exposure to inappropriate content) and poor child outcomes. Research shows that exposure to screen media and externalizing behavior problems in young children are linked. Externalizing behavior problems also present a significant barrier to parents attempting to adhere to screen media use recommendations. Despite these public health concerns, screen media use interventions have not yet specifically targeted children with externalizing behavior problems. To address this need, the investigators propose to explore a novel approach to intervening around screen time, by adapting a behavioral parenting intervention designed for parents of children with externalizing behavior problems to integrate content around screen time. Leveraging an existing evidence-based parenting intervention will allow for the intervention to target parenting generally, as well as screen time specific parenting, without requiring additional resources. This study will focus on adapting a group-based parenting intervention, the School Readiness Parenting Program (SRPP). The SRPP is an 8-week parenting intervention based on a group Parent-Child Interaction Therapy model. In total, 55 parents of preschool-aged children with externalizing behavior problems will be recruited. Following a development phase, the investigators will conduct a small open trial (n = 15) to assess the feasibility of the screen time adapted intervention and families' satisfaction and response to treatment. At this phase, the investigators will also pilot a multimodal method of tracking child screen use using objective data from mobile devices and parent-completed media use logs. Upon making modifications based on results of the open trial and feedback from an external advisory panel of experts and community stakeholders, a pilot randomized controlled trial (n = 40) will follow. Parents will be randomly assigned to receive either the screen time adapted SRPP (n = 20) or the original SRPP (n = 20) program. Assessment measures will be completed at prettest, posttest, and at a 1 month follow up. The investigators will examine feasibility and acceptability of the screen time adapted intervention in the randomized controlled trial. The investigators will also examine children's screen use patterns, including overall screen time, proportion of screen time that is educational, and frequency of parent-child co-use of screen media. In an exploratory fashion, the investigators will examine the effect of the intervention on child externalizing behavior problems.

ELIGIBILITY:
Inclusion Criteria:

* eligible child who is 54 to 66 months old at Spring intake (i.e. will be entering Kindergarten after the summer)
* parent-reported externalizing behavior problems on the Kiddie-Disruptive Behavior Disorder Schedule (parent report) or the Disruptive Behavior Disorder Rating Scale (teacher report) that meet criteria for a disruptive behavior disorder diagnosis
* child general cognitive ability score 70 or above on the Differential Abilities Scales-II, - caregiver willing and able to attend weekly parent groups conducted in English.

Exclusion Criteria:

* Families with children with major sensory impairments (e.g., deafness, blindness) or severe problems that impair mobility (e.g., cerebral palsy)are excluded.

Ages: 54 Months to 66 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
A controlled access approach, using a robust system to review requests and provide secure access to de-identified data, will be utilized.
Supporting Information: Study Protocol
Time Frame: Deidentified data for the entire database will be made available for data sharing after the main findings from the final dataset have been accepted for publication.
Access Criteria: Users will be provided with the data under a data-sharing agreement which specifies that: (1) data will be used only for research purposes; (2) data will be stored confidentially and securely; and (3) data will be destroyed after analyses are completed. PI Bagner and collaborators will identify where the data will be available and how to access the data in any publications and presentations using these data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for the open trial (n = 10) and the pilot RCT (n = 34) were recruited from families attending Summer Academy, an 8-week summer camp for preschoolers with externalizing behavior.
Pre-assignment Details: For the open trial period, 28 participants were assessed for eligibility, and 10 were eligible and elected to participate (all assigned to Screen media adapted School Readiness Parenting Program). For the RCT period 142 participants were assessed for eligibility, and of these, 34 met criteria and were randomized to treatment. Participants in the open trial did not participate in the RCT.
Period: Open Trial
Arm/Group | Screen Media Adapted School Readiness Parenting Program | Original School Readiness Parenting Program
Started | 10 | 0
Received Intervention | 10 | 0
Post-test | 10 | 0
Completed | 10 | 0
Not Completed | 0 | 0
Period: Pilot Randomized Controlled Trial
Arm/Group | Screen Media Adapted School Readiness Parenting Program | Original School Readiness Parenting Program
Started | 18 | 16
Received Intervention | 16 | 15
Post-test | 16 | 15
Completed | 15 | 15
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline participants include participants in the open trial in Year 1, who recieved the adapted intervention, and participants in the RCT in year 2, who were randomized to receive either the adapted or the standard intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Screen Media Adapted School Readiness Parenting Program | Original School Readiness Parenting Program | Total
Number analyzed (Participants) | 26 | 15 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] — Caregiver age in years Population: 3 participants discontinued participation before the intervention was delivered and were not included in the analyses.
  years | 34.26 (6.168) | 33.21 (7.71) | 33.85 (6.59)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 participants discontinued participation before intervention was delivered, and were excluded from analyses
  Participants
    Female | 23 | 4 | 27
    Male | 3 | 11 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 participants discontinued participation before intervention was complete and were not included in analyses
  Participants
    Hispanic or Latino | 4 | 5 | 9
    Not Hispanic or Latino | 22 | 10 | 32
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 participants discontinued participation before the intervention was delivered, and were not included in analyses
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 18 | 9 | 27
    White | 7 | 5 | 12
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 0 | 0 | 0
Child screen media use (average weekend day) [Mean (Standard Deviation); unit: minutes per day] — Population: 3 participants discontinued participation before receiving the intervention, and were not included in analyses
  minutes per day | 256.15 (152.35) | 226.00 (207.51) | 245.12 (172.61)
Child screen media use (average weekday) [Mean (Standard Deviation); unit: minutes per day] — Population: 3 participants discontinued participation before receiving the intervention, and were not included in analyses
  minutes per day | 190.57 (148.27) | 242.67 (156.35) | 209.63 (151.47)
Child screen media use (proportion educational) [Mean (Standard Deviation); unit: proportion of total screen media use] — Caregivers reported the proportion of their child's screen media use that was educational Population: 3 participants discontinued participation before receiving the intervention, and were not included in analyses
  proportion of total screen media use | .33 (.21) | .39 (.23) | .35 (.22)
Perceived Parental Efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — Parents' perceived efficacy in managing children's screen time was assessed using the Perceived Parental Efficacy subscale of the Parent Perceptions of Technology Scale (PPTS), which assesses parents' self-efficacy in using electronic media and managing children's screen time (e.g., "I won't bother setting parental controls or passwords because my kids will "hack" around them."). The 5 items were rated on a Likert scale from 1 (strongly disagree) to 5 (strongly agree). Population: 3 participants discontinued participation before receiving the intervention, and were not included in analyses
  units on a scale | 4.11 (.58) | 4.34 (.64) | 4.20 (.61)
Technology-related Parenting Scale [Mean (Standard Deviation); unit: units on a scale] — 4 items from the Technology-related Parenting Scale were used to assess parents' use of rules and limit-setting (e.g., "I set limits on the amount of time") for children's technology use on a 3-point scale from 0 (not true) to 2 (very true). Population: 3 participants discontinued participation before receiving the intervention, and were not included in analyses
  units on a scale | 1.36 (.62) | 1.45 (.42) | 1.39 (.55)

OUTCOME MEASURES:

1. Primary Outcome: Child Screen Media Use (Time)
Description: Child screen media use will be measured with parent-reported data on screen use duration (including TV and other screen devices) and content. The outcome variable will be total screen use per weekend day.
Time Frame: Change from baseline (week 0) to posttest (week 8) and follow-up (week 16)
Population: Analysis population includes participants in the open trial who attended more than haft of the groups sessions (n = 7) as well as participants in the randomized trial. All participants in the randomized trial who began the intervention program were included in the analyses (n = 31). One participant in the pilot RCT was lost to follow up at the follow up (week 16) time point.
Measure: Mean (Standard Deviation); unit: minutes per weekend day
Arm/Group | Screen Media Adapted School Readiness Parenting Program | Original School Readiness Parenting Program
Number analyzed (Participants) | 23 | 15
minutes per weekend day
  Open Trial - Baseline: number analyzed (Participants) | 7 | 0
  Open Trial - Baseline | 210.00 (89.58) |
  Open Trial - Posttest: number analyzed (Participants) | 7 | 0
  Open Trial - Posttest | 267.86 (124.76) |
  Open Trial - Follow-up: number analyzed (Participants) | 7 | 0
  Open Trial - Follow-up | 163.57 (100.57) |
  Pilot RCT - Baseline: number analyzed (Participants) | 16 | 15
  Pilot RCT - Baseline | 290.00 (177.29) | 226.00 (207.51)
  Pilot RCT - Posttest: number analyzed (Participants) | 16 | 15
  Pilot RCT - Posttest | 155.94 (76.38) | 225.00 (210.56)
  Pilot RCT - Follow-Up: number analyzed (Participants) | 15 | 15
  Pilot RCT - Follow-Up | 160.00 (80.29) | 198.67 (183.08)
Statistical Analysis 1: Comparison: Screen Media Adapted School Readiness Parenting Program; Preliminary pre-post outcome analysis for the open trial (n = 7). The analysis was a paired samples t-test comparing baseline (week 0) to posttest (week 8) scores; Test type: Other; p = .29, t-test, 2 sided
Statistical Analysis 2: Comparison: Screen Media Adapted School Readiness Parenting Program; Preliminary outcome analysis for the open trial (n = 7). The analysis was a paired samples t-test comparing baseline(week 0) to follow-up (week 16) scores; Test type: Other; p = .34, t-test, 2 sided
Statistical Analysis 3: Comparison: Screen Media Adapted School Readiness Parenting Program vs Original School Readiness Parenting Program; ANCOVA analysis for the pilot RCT, comparing the outcome variable at posttest (Week 8) between the two groups, with pretest (baseline) scores, annual household income and household size (to approximate income-to-needs ratio), caregiver education, and child externalizing behavior as covariates; Test type: Superiority; p = .02, ANCOVA
Statistical Analysis 4: Comparison: Screen Media Adapted School Readiness Parenting Program vs Original School Readiness Parenting Program; ANCOVA analysis for the pilot RCT, comparing the outcome variable at follow-up (Week 16) between the two groups, with pretest (baseline) scores, annual household income and household size (to approximate income-to-needs ratio), caregiver education, and child externalizing behavior as covariates; Test type: Superiority; p = .04, ANCOVA

2. Primary Outcome: Child Screen Media Use (Proportion Educational)
Description: The proportion of child screen media use that parents report is educational.
Time Frame: Change from baseline (week 0) to posttest (week 8) and follow-up (week 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of total media content
Arm/Group | Screen Media Adapted School Readiness Parenting Program | Original School Readiness Parenting Program
Number analyzed (Participants) | 23 | 15
proportion of total media content
  Open Trial - Baseline: number analyzed (Participants) | 7 | 0
  Open Trial - Baseline | .36 (.15) |
  Open Trial - Posttest: number analyzed (Participants) | 7 | 0
  Open Trial - Posttest | .37 (.17) |
  Open trial - Follow-Up: number analyzed (Participants) | 7 | 0
  Open trial - Follow-Up | .34 (.16) |
  Pilot RCT - Baseline: number analyzed (Participants) | 16 | 15
  Pilot RCT - Baseline | .34 (.22) | .39 (.23)
  Pilot RCT - Posttest: number analyzed (Participants) | 16 | 15
  Pilot RCT - Posttest | .38 (.16) | .40 (.21)
  Pilot RCT - Follow-Up: number analyzed (Participants) | 15 | 15
  Pilot RCT - Follow-Up | .41 (.18) | .40 (.22)
Statistical Analysis 1: Comparison: Screen Media Adapted School Readiness Parenting Program; Preliminary outcome analysis for the open trial (n = 7). The analysis was a paired samples t-test comparing baseline (week 0) to posttest (week 8) scores; Test type: Other; p = .88, t-test, 2 sided
Statistical Analysis 2: Comparison: Screen Media Adapted School Readiness Parenting Program; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = .87, t-test, 2 sided
Statistical Analysis 3: Comparison: Screen Media Adapted School Readiness Parenting Program vs Original School Readiness Parenting Program; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = .10, ANCOVA
Statistical Analysis 4: Comparison: Screen Media Adapted School Readiness Parenting Program vs Original School Readiness Parenting Program; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = .90, ANCOVA

3. Primary Outcome: Treatment Attitude Inventory (TAI)
Description: The TAI is a parent-report measure that assesses parent satisfaction with treatment. Test-retest reliability over 4 months and correlations between the TAI and both parent-rating scales and observational measures of treatment change have been demonstrated. The TAI total score will be administered to assess parent satisfaction with the intervention. The minimum value is 0 and the maximum is 50, with higher scores indicating better satisfaction.
Time Frame: Posttest (Week 8)
Population: Analysis population includes participants in the open trial (n = 10) as well as participants in the randomized trial. All participants in the randomized trial who began the intervention program were included in the analyses (n = 31).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Screen Media Adapted School Readiness Parenting Program | Original School Readiness Parenting Program
Number analyzed (Participants) | 26 | 15
units on a scale
  Open trial - Posttest: number analyzed (Participants) | 10 | 0
  Open trial - Posttest | 44.60 (5.37) |
  Pilot RCT - Posttest: number analyzed (Participants) | 16 | 15
  Pilot RCT - Posttest | 45.19 (4.75) | 45.64 (4.92)
Statistical Analysis 1: Comparison: Screen Media Adapted School Readiness Parenting Program vs Original School Readiness Parenting Program; T-test analysis for the pilot RCT, comparing the outcome variable at posttest (Week 8) between the two groups; Test type: Equivalence — Analysis to test whether groups had equivalent levels of satisfaction with treatment (defined as the groups not being significantly different at the level of p<.05); p = .80, t-test, 2 sided

4. Primary Outcome: Perceived Parental Efficacy Scale
Description: Parents' perceived efficacy in managing children's screen time will be assessed using the Perceived Parental Efficacy subscale of the Parent Perceptions of Technology Scale (PPTS), which assesses parents' self-efficacy in using electronic media and managing children's screen time (e.g., "I won't bother setting parental controls or passwords because my kids will "hack" around them."). The 5 items are rated on a Likert scale from 1 (strongly disagree) to 5 (strongly agree). Items were reverse scored and averaged to create the overall scale score, with higher scores meaning better perceived efficacy.
Time Frame: Change from baseline (week 0) to posttest (week 8) and follow-up (week 16).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Screen Media Adapted School Readiness Parenting Program | Original School Readiness Parenting Program
Number analyzed (Participants) | 23 | 15
units on a scale
  Open Trial - Baseline: number analyzed (Participants) | 7 | 0
  Open Trial - Baseline | 4.12 (.71) |
  Open Trial - Posttest: number analyzed (Participants) | 7 | 0
  Open Trial - Posttest | 4.36 (.81) |
  Open Trial - Follow-Up: number analyzed (Participants) | 7 | 0
  Open Trial - Follow-Up | 4.62 (.51) |
  Pilot RCT - Baseline: number analyzed (Participants) | 16 | 15
  Pilot RCT - Baseline | 4.05 (.56) | 4.34 (.64)
  Pilot RCT - Posttest: number analyzed (Participants) | 16 | 15
  Pilot RCT - Posttest | 4.23 (.70) | 4.50 (.55)
  Pilot RCT - Follow- Up: number analyzed (Participants) | 15 | 15
  Pilot RCT - Follow- Up | 4.11 (.61) | 4.53 (.57)
Statistical Analysis 1: Comparison: Screen Media Adapted School Readiness Parenting Program; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = .35, t-test, 2 sided
Statistical Analysis 2: Comparison: Screen Media Adapted School Readiness Parenting Program; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = .049, t-test, 2 sided
Statistical Analysis 3: Comparison: Screen Media Adapted School Readiness Parenting Program vs Original School Readiness Parenting Program; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = .45, ANCOVA
Statistical Analysis 4: Comparison: Screen Media Adapted School Readiness Parenting Program vs Original School Readiness Parenting Program; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = .20, ANCOVA

5. Primary Outcome: Technology-related Parenting Scale
Description: The Technology-related Parenting Scale is an 8-item self-report survey assessing parents' use of rules (e.g., "I set limits on the amount of time") and enforcement strategies ("I use passwords on these devices") for children's technology use on a 3-point scale from 0 (not true) to 2 (very true). Items will be averaged to create an overall score, with higher scores meaning more limit setting.
Time Frame: Change from baseline (week 0) to posttest (week 8) and follow-up (week 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Screen Media Adapted School Readiness Parenting Program | Original School Readiness Parenting Program
Number analyzed (Participants) | 23 | 15
units on a scale
  Open Trial - Baseline: number analyzed (Participants) | 7 | 0
  Open Trial - Baseline | .92 (.71) |
  Open Trial -Posttest: number analyzed (Participants) | 7 | 0
  Open Trial -Posttest | 1.71 (.30) |
  Open Trial - Follow-Up: number analyzed (Participants) | 7 | 0
  Open Trial - Follow-Up | 1.59 (.70) |
  Pilot RCT - Baseline: number analyzed (Participants) | 16 | 15
  Pilot RCT - Baseline | 1.48 (.56) | 1.45 (.42)
  Pilot RCT - Posttest: number analyzed (Participants) | 16 | 15
  Pilot RCT - Posttest | 1.70 (.42) | 1.76 (.27)
  Pilot RCT - Follow-Up: number analyzed (Participants) | 15 | 15
  Pilot RCT - Follow-Up | 1.66 (.41) | 1.76 (.43)
Statistical Analysis 1: Comparison: Screen Media Adapted School Readiness Parenting Program; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = .006, t-test, 2 sided
Statistical Analysis 2: Comparison: Screen Media Adapted School Readiness Parenting Program; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = .011, t-test, 2 sided
Statistical Analysis 3: Comparison: Screen Media Adapted School Readiness Parenting Program vs Original School Readiness Parenting Program; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = .22, ANCOVA
Statistical Analysis 4: Comparison: Screen Media Adapted School Readiness Parenting Program vs Original School Readiness Parenting Program; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = .25, ANCOVA

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Screen Media Adapted School Readiness Parenting Program | Original School Readiness Parenting Program
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/15
Other Adverse Events (participants affected / at risk) | 0/26 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT05287685/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT05287685/ICF_001.pdf